CLINICAL TRIAL: NCT04554108
Title: Acute Non-severe Osteomyelitis in Children - Outpatient Management Strategy With Oral Antibiotic Therapy Compared to a Standard Strategy With Conventional Hospitalization and Intravenous Antibiotic Therapy: a Randomized Open-label Non-inferiority Study With Bayesian and Medical-economic Analyses.
Acronym: POOMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP180672; 2019-003522-25 (EudraCT Number)
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Osteomyelitis
MeSH Terms: conditions — Osteomyelitis

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial of non inferiority, with active control, in open multicenter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous antibiotic treatment (Active Comparator): Intravenous antibiotic treatment started during an initial hospitalization of 3 days, with continuation of oral antibiotic therapy at home for a total duration of antibiotic therapy of 3 weeks
  Interventions: Other: therapeutic strategy
- oral antibiotic treatment (Experimental): Oral antibiotic treatment started in hospital then continued at home for a total duration of 3 weeks of antibiotic therapy
  Interventions: Other: therapeutic strategy

INTERVENTIONS:
Other: therapeutic strategy — Outpatient management strategy of acute non-severe osteomyelitis in children with oral antibiotic therapy compared to a standard strategy with conventional hospitalization and intravenous antibiotic therapy

SUMMARY:
The incidence of bone and joint infections (BJI) in children (osteomyelitis, septic arthritis and spondylodiscitis) is 22 per 100,000 children in France. Every year, 3,000 children are hospitalized for BJI, 46% of whom are hospitalized for osteomyelitis. The clinical pictures of BJI are varied: some are severe from the outset; others are non-severe, such as BJIs in Kingella kingae, which are most common in children between the ages of 6 months and 5 years. Currently, the management of children's BJI, regardless of their severity, involves initial hospitalization to start intravenous antibiotic therapy. This non-inferiority trial evaluates, in children with acute osteomyelitis with no severity criteria, less invasive outpatient management with an oral antibiotic treatment given at the outset compared to standard management.

Main objective : Demonstrate the non-inferiority of an ambulatory management strategy versus a standard strategy involving hospitalization on complete recovery without relapse at 6 months after an episode of acute osteomyelitis in children aged 1-4 years without severity criteria.

Primary endpoint: Complete cure without relapse at 6 months defined by the absence of clinical signs of osteomyelitis at 6 months AND the absence of secondary septic complications (septic arthritis, periosteal abscess) before the end of antibiotic therapy AND the absence of relapse or rehospitalization for osteomyelitis related to the initial infection. This criterion will be assessed blindly by an adjudication committee.

Randomized controlled trial of non inferiority, with active control, in open multi-center.

The control or experimental arm allocation (1:1 ratio) will be open-label of the physician, patient and parents. This is a PROBE study: The evaluation of the main judgment criterion will be carried out blindly by an adjudication committee.

DETAILED DESCRIPTION:
The incidence of bone and joint infections (BJI) in children (osteomyelitis, septic arthritis and spondylodiscitis) is 22 per 100,000 children in France. Every year, 3,000 children are hospitalized for BJI, 46% of whom are hospitalized for osteomyelitis. The clinical pictures of BJI are varied: some are severe from the outset; others are non-severe, such as BJIs in Kingella kingae, which are most common in children between the ages of 6 months and 5 years. Currently, the management of children's BJI, regardless of their severity, involves initial hospitalization to start intravenous antibiotic therapy. This non-inferiority trial evaluates, in children with acute osteomyelitis with no severity criteria, less invasive outpatient management with an oral antibiotic treatment given at the outset compared to standard management.

Main objective : Demonstrate the non-inferiority of an ambulatory management strategy versus a standard strategy involving hospitalization on complete recovery without relapse at 6 months after an episode of acute osteomyelitis in children aged 1-4 years without severity criteria.

Primary endpoint: Complete cure without relapse at 6 months defined by the absence of clinical signs of osteomyelitis at 6 months AND the absence of secondary septic complications (septic arthritis, periosteal abscess) before the end of antibiotic therapy AND the absence of relapse or rehospitalization for osteomyelitis related to the initial infection. This criterion will be assessed blindly by an adjudication committee.

Randomized controlled trial of non inferiority, with active control, in open multi-center.

The control or experimental arm allocation (1:1 ratio) will be open-label of the physician, patient and parents. This is a PROBE study: The evaluation of the main judgment criterion will be carried out blindly by an adjudication committee.

ELIGIBILITY:
Inclusion Criteria:

Child ≥ 1 year and 4 years old ;

* First episode of acute osteomyelitis suspected on clinical grounds (acute functional impotence (<15 days) most often associated with fever) and confirmed in the first days of treatment by bone scan or MRI.
* Absence of severity criteria :

  * Fever < 39°C
  * AND absence of sepsis (absence of hemodynamic disorders, respiratory disorders, consciousness disorders)
  * AND absence of periosteal abscess or associated arthritis or deep vein thrombosis
  * AND absence of scarlatiniform rash (no gap of healthy skin)
  * AND CRP < 50 mg/ml
  * AND normal initial bone radiograph (or simple soft tissue thickening).

Exclusion Criteria:

* Multifocal osteoarticular infections
* Sickle cell or immunocompromised patients
* Antibiotic treatment in progress or within 48 hours prior to the emergency room visit
* History of severe beta-lactam allergy (anaphylactic shock, angioedema)
* Digestive problems (vomiting or diarrhea)
* Refusal of parents to participate
* Parents (children) not affiliated to social security or without CMU
* Parents who do not speak French
* Participation in another intervention research protocol

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Complete recovery without relapse at 6 months | 6 months
  Complete recovery without relapse defined by the absence of clinical signs of osteomyelitis (absence of pain, fever, swelling & heat of any limb, biological inflammatory signs, relapse or hospitalisation AND the absence of secondary septic complications (septic arthritis, sub-periosteal abscess)

CONTACTS AND LOCATIONS:
Overall Officials: Mathie LORROT, MD PhD, Principal Investigator — APHP
Locations (1):
- Trousseau Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No